CLINICAL TRIAL: NCT01995604
Title: A Single Center, Double Blinded, Placebo Controlled, Randomized, Split Face Study to Evaluate the Efficacy of dHACM (Dehydrated Human Amnion Chorion Membrane) for Recovery After Fractionated Ablative CO2 Laser Resurfacing of the Face
Brief Title: Dehydrated Human Amnion/Chorion Membrane (dHACM) for Recovery After Fractionated Ablative CO2 Laser Resurfacing of the Face
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFLR001
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Scarring
MeSH Terms: conditions — Cicatrix | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dHACM (Experimental): UltraPulse laser therapy with application of dHACM
  Interventions: Other: Application of dHACM
- Sterile 0.9% Saline Solution (Placebo Comparator): UltraPulse laser therapy with application of Sterile 0.9% Saline Solution
  Interventions: Other: Application of Sterile 0.9% Saline Solution

INTERVENTIONS:
Other: Application of Sterile 0.9% Saline Solution — Application of Sterile 0.9% Saline Solution to half of face after UltraPulse laser therapy.
  Arms: Sterile 0.9% Saline Solution
Other: Application of dHACM — Application of dHACM to half of face after UltraPulse laser therapy.
  Arms: dHACM

SUMMARY:
The purpose of this study is to evaluate the efficacy of dHACM (Dehydrated Human Amnion Chorion Membrane) for reducing time to healing when used in post-laser recovery following ActiveFX™ and DeepFx™ fractionated ablative CO2 laser resurfacing of the face.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects in good general health greater than 18 years of age
2. Must be willing to agree to all terms of the protocol and provide a completed and signed informed consent, HIPAA and photography release forms
3. Subjects planning to undergo fractionated ablative CO2 laser resurfacing to the full face
4. Subject of either Fitzpatrick Skin Types I, II or III

   * For female subjects of childbearing potential, they must have had a regular menstrual cycle prior to study entry and is willing to use an acceptable form of birth control during the entire course of the study. All systemic birth control measures must be in consistent use at least 30 days prior to entry into the study. A female is considered NOT to be of childbearing potential if she is postmenopausal for at least one (1) year, without a uterus and/or both ovaries, or has had a bilateral tubal ligation. Acceptable methods of birth control are: oral contraceptives, contraceptive patches/rings/implants Norplant, Depo-Provera, double-barrier methods (e.g. condoms and spermicide), abstinence and vasectomies of the partner.
5. Negative urine pregnancy test results at the time of study entry for females of childbearing potential, if applicable
6. Must be willing to comply with study instructions and complete the entire course of the study

Exclusion Criteria:

1. Any uncontrolled systemic disease that is not yet stabilized for at least one (1) year
2. A significant history or current evidence of a medical, psychological or other disorder that, in the investigator's opinion, would interfere with the objectives of the study
3. Recently excessive exposure to sunlight or artificial UV light (e.g.: use of tanning beds/booths and/or sunbathing) or expectations of tanning during the time of the study or has used self-tanner within 7 days of study entry
4. History of or the presence of any skin condition/disease that might interfere with the diagnosis or evaluation of study parameters (i.e., atopic dermatitis, eczema, psoriasis, seborrheic dermatitis)
5. Active bacterial, fungal, or viral infection
6. History of Herpes Simplex Virus to the facial and/or perioral areas
7. Known allergies or sensitivities to benzocaine, lidocaine, tetracaine, PABA (para-aminobenzoic acid), or other local anesthetics of the amide or ester family
8. Known allergies to gentamicin and/or streptomycin
9. Receiving any topical products containing alpha-hydroxy acids, salicylic acid, and Vitamins C or E (including derivatives of Vitamins C or E) on the face within 14 days prior to or during the study period, other than the ingredients of the study products
10. Receiving and/or has had a microdermabrasion (light or medium skin peel) treatment on their face within 30 days prior to or during the study period
11. Using any topical tretinoin product or derivative on their face within 12 weeks prior to or during the study period
12. Receiving a chemical peel, any systemic steroids, a non-ablative laser, light or radio frequency treatment and/or has had a Dermabrasion (deep skin peel) or ablative laser treatments on their face must have discontinued the drug/treatment and/or had the procedure at least 3 months prior to entering the study
13. History of keloids or hypertrophic scars
14. Use of systemic retinoids, prescription or over-the-counter grade within the past year
15. A female subject who is pregnant, nursing an infant or planning a pregnancy during the study
16. Current participation or completed participation of a clinical research study for an investigational drug or device within 30 days prior to the start of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The time to healing for both groups will be assessed as defined by appearance and 100% epithelialization. | Day 30

SECONDARY OUTCOMES:
Erythema, edema, crusting, and exudate will be compared between both groups. | 30 Days

OTHER OUTCOMES:
Pain Reduction | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Mitchel P Goldman, MD, Principal Investigator — Dermatology Cosmetic Laser Medical Associates of La Jolla, Inc.
Locations (1):
- Dermatology Cosmetic Laser Medical Associates of LaJolla, Inc., San Diego, California, United States